CLINICAL TRIAL: NCT01762514
Title: A Multi-institutional, Randomized Parallel Controlled, Phase II Clinical Trial on Comparison of Effectiveness and Safeness of Amifostine Every-other-day Regimen and Everyday Regimen From Monday to Friday
Brief Title: A Phase II Clinical Trial on Comparison of Effectiveness and Safeness of Different Amifostine Regimens
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Dalian Merro Pharmaceutical Co. Ltd (Unknown)
Responsible Party: Principal Investigator, Yun-fei Xia, Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMF-BYA-02
Record Dates: First submitted 2012-12-22; First posted 2013-01-07 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Nasopharyngeal Neoplasms; Salivary Gland Diseases; Bone Marrow Diseases; Mucositis
Keywords: Nasopharyngeal carcinoma; Amifostine; Myelosuppression; Xerostomia; Mucositis
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Salivary Gland Diseases; Bone Marrow Diseases; Mucositis; Nasopharyngeal Carcinoma; Xerostomia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Program I (No Intervention): Patients with American Joint Cancer Committee/Union Internationale Contre le Cancer (UICC/AJCC) 2010 Stage I and II; Radiotherapy applied
- Program II (Experimental): Patients with UICC/AJCC 2010 Stage I and II; Radiotherapy applied; Amifostine every-other-day regimen
  Interventions: Drug: Amifostine every-other-day regimen
- Program III (Active Comparator): Patients with UICC/AJCC 2010 Stage I and II; Radiotherapy applied; Amifostine everyday regimen
  Interventions: Drug: Amifostine everyday regimen
- Program IV (No Intervention): Patients with UICC/AJCC 2010 Stage III, IVa and IVb; Concurrent chemoradiotherapy applied
- Program V (Experimental): Patients with UICC/AJCC 2010 Stage III, IVa and IVb; Concurrent chemoradiotherapy applied; Amifostine every-other-day regimen
  Interventions: Drug: Amifostine every-other-day regimen
- Program VI (Active Comparator): Patients with UICC/AJCC 2010 Stage III, IVa and IVb; Concurrent chemoradiotherapy applied; Amifostine everyday regimen
  Interventions: Drug: Amifostine everyday regimen

INTERVENTIONS:
Drug: Amifostine every-other-day regimen — Amifostine 400mg/d, every-other-day regimen from Monday to Friday, every week repetition during radiotherapy
  Other Names: Amifostine administered 3 times per week regimen
  Arms: Program II; Program V
Drug: Amifostine everyday regimen — Amifostine 400mg/d, everyday regimen from Monday to Friday, every week repetition during radiotherapy
  Other Names: Amifostine administered 5 times per week regimen
  Arms: Program III; Program VI

SUMMARY:
RATIONALE

* Radiotherapy is the primary therapeutic strategy for nasopharyngeal carcinoma.
* Radiotherapy may cause adverse effect such as xerostomia and mucositis.
* Amifostine has the ability of protecting the normal tissue but also has some side effects.

PURPOSE

* This phase II trial is to study the protecting effect and safety of different Amifostine regimens in patients with nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
RATIONALE: Nasopharyngeal carcinoma is a kind of malignant tumor which is treated primarily by radiation therapy. This therapeutic strategy often causes adverse effects such as dysfunction of salivary gland and lesion of oral mucosa. With concurrent chemotherapy, it may also cause toxicity to kidney, bone marrow, and other organs or tissues. When administered prior to chemoradiotherapy, Amifostine has been proved to has the ability of protecting the normal from these adverse effects so as to improve the patient tolerance. However, there are also some side effects of Amifostine itself, such as nausea, vomiting and hypotension, especially when high dose is applied.

PURPOSE: This phase II randomized controlled trial is to study the protecting effect and its safety of Amifostine every-other-day regimen compared with standard everyday regimen on adverse effects such as myelosuppression, xerostomia and mucositis, in patients with nasopharyngeal carcinoma Stage T1-T4, N0-N3, M0 and undergoing concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal cancer patients diagnosed by pathology or cytology
* UICC/AJCC 2010 Stage T1-4 N0-3 M0
* Male or female patients with age between 18 and 75 years old
* Karnofsky Performance Scores ≥ 60
* Expected survival ≥ 3 months
* Without dysfunction of heart, lung, liver, kidney and hematopoiesis
* No previous allergic reaction to the drug

Exclusion Criteria:

* History of alcohol or drug abuse within 3 months
* Pregnant or lactating women
* Currently under treatment with other similar drugs
* Anti-hypertension drugs applied in less than 24 hours
* Severe hypocalcemia
* Dysfunction of heart, lung, liver, kidney or hematopoiesis
* Severe neurological, mental or endocrine diseases
* Previous allergic reaction to the drug
* Patients participated in clinical trials of other drugs within last 3 months
* Other unsuitable reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Effect on improving myelosuppression | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
  Severity of myelosuppression is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria.
Effect on improving xerostomia | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
  Severity of xerostomia is evaluated on basis of CTCAE 4.0 criteria.
Effect on improving mucositis | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
  Severity of mucositis is evaluated on basis of CTCAE 4.0 criteria.

SECONDARY OUTCOMES:
Effect on improving Quality of Life (QOL). | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
Effect on improving Karnofsky Performance Scores (KPS) | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
Incidence and severity of Nausea | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
  One of the adverse effects of Amifostine.
Incidence and severity of Vomiting | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
  One of the adverse effects of Amifostine.
Incidence and severity of Hypotension | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
  One of the adverse effects of Amifostine.
Incidence and severity of Hypocalcemia | One week before radiotherapy; Once a week during radiotherapy, up to 7 weeks; Three months after radiotherapy
  One of the adverse effects of Amifostine.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, Prof., Principal Investigator — Department of Radiation Oncology, Sun Yat-Sen University Cancer Center
Locations (7):
- China (7):
  - The Main Guangzhou Hospital of the Guangzhou Military Region, Guangzhou, Guangdong
  - Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The Affiliated Cancer Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong
  - Guangdong Provincial Hospital Of Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong
  - The Second Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangdong Second People's Hospital, Guangzhou, Guangdong

REFERENCES:
- [Derived] Liu Y, Shi H, Huang S, Chen X, Zhou H, Chang H, Xia Y, Wang G, Yang X. Early prediction of acute xerostomia during radiation therapy for nasopharyngeal cancer based on delta radiomics from CT images. Quant Imaging Med Surg. 2019 Jul;9(7):1288-1302. doi: 10.21037/qims.2019.07.08. PMID 31448214
- [Derived] Chang H, Yi W, Wang X, Tao Y, Yang X, Chen C, Zhang W, Zhou S, Liu S, Li X, Ding S, Li J, Li G, Shao X, Liu Y, Song W, Xia Y. Effectiveness and safety of different amifostine regimens: Preliminary results of a phase II multicenter randomized controlled trial. Chin J Cancer Res. 2018 Jun;30(3):307-314. doi: 10.21147/j.issn.1000-9604.2018.03.03. PMID 30046225